CLINICAL TRIAL: NCT05990465
Title: Phase I Study of LV20.19 CAR T-cells in Combination With Pirtobrutinib for Relapsed, Refractory B-cell Malignancies
Brief Title: LV20.19 CAR T-Cells in Combination With Pirtobrutinib for Relapsed, Refractory B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nirav Shah, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00050826
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Non Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Burkitt Lymphoma
Keywords: CAR-T; Chimeric antigen receptor T-cell therapy; CAR Therapy; Pirtobrutinib; B Cells; BTK inhibitor; Bruton's tyrosine kinase
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Burkitt Lymphoma | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pirtobrutinib and CAR T Cells (Experimental): Pirtobrutinib is an oral agent. LV20.19 CAR T cells will be administered either fresh or thawed after cryopreservation by IV injection.
  Interventions: Drug: Pirtobrutinib; Drug: LV20.19 CAR T cells

INTERVENTIONS:
Drug: Pirtobrutinib — Pirtobrutinib will be administered at 200 mg/day orally starting at least 14 days prior to apheresis as bridging until the start of lymphodepletion and restarted between day 28-120 for up to one year as maintenance post cell infusion.
  Other Names: Jaypirca; LOXO-305
Drug: LV20.19 CAR T cells — Subjects will receive a dose of 2.5x10^6 CAR-T cells/kg as a previously identified safe in a Phase 1 protocol at the Medical College of Wisconsin.

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study designed to evaluate the safety and efficacy of LV20.19 CAR -T cells with pirtobrutinib bridging and maintenance in adult patients with B cell malignancies that have failed prior therapies.

DETAILED DESCRIPTION:
This is the first study to evaluate the safety and impact of the combination of pirtobrutinib and LV20.19 CAR-T cells.

Pirtobrutinib is a first-in-class non-covalent Bruton's tyrosine kinase (BTK) inhibitor. The safe dose of this agent has been identified the BRUIN study as 200 mg daily administered as an oral agent. As a single agent, the toxicity profile has been favorable and does not overlap with other covalent BTK inhibitors with minimal cardiotoxicity and bleeding complications.

ELIGIBILITY:
To facilitate rapid start of pirtobrutinib, there will be separate inclusion/exclusion for pirtobrutinib and LV20.19 CAR T-cells in addition to the general inclusion as outlined below.

General inclusion criteria for trial:

1. Patients must be aged ≥18 years and <81 years with relapsed or refractory B-cell non-Hodgkin Lymphoma (NHL).
2. Diagnosis of relapsed or refractory B-cell NHL including Follicular Lymphoma, Marginal Zone Lymphoma (splenic, nodal, extranodal), Mantle Cell Lymphoma, Burkitt Lymphoma and DLBCL with associated subtypes (aggressive B-cell lymphoma, high grade B-cell lymphoma, T-cell/histocyte rich B-cell lymphoma, primary mediastinal B-cell lymphoma, Epstein-Barr virus-positive (EBV)+ diffuse large B-cell lymphoma, transformed lymphoma such as transformed follicular or marginal zone, and Richter's transformation).
3. Disease specific criteria as follows:

   1. DLBCL and associated subtypes (listed above)

   i. Must have received Rituximab or another cluster of differentiation 20 (CD20) antibody with combination anthracycline based chemotherapy regimen and have ONE of the following:

<!-- -->

1. Primary refractory lymphoma or early relapse ≤6 months after one line of therapy.
2. For relapse >6.00 months, failure of two different chemotherapy regimens appropriate for their disease and be ineligible to receive autologous transplant.

ii. Relapse post-autologous transplant. iii. Relapse post-allogeneic transplant. iv. Relapse post-CAR T-cell therapy (maximum 2 patients allowed with this designation).

b. Mantle Cell Lymphoma

i. Must have received Rituximab or another CD 20 antibody with one chemotherapy regimen appropriate for this disease (bendamustine or cytarabine, or anthracycline based treatment) and have ONE of the following:

1. Relapsed disease after two lines of cytotoxic chemotherapy including administration of anti-CD20 antibody.
2. Progressive disease after ≥second line BTK inhibitor.
3. Relapse post-autologous transplant.
4. Relapse post-allogeneic transplant.

   c. Marginal Zone Lymphoma and Follicular Lymphoma

   i. Must have received Rituximab or another CD20 antibody with chemotherapy regimen appropriate for the disease and have ONE of the following:

<!-- -->

1. Relapsed disease after two lines of therapy including administration of anti-CD20 antibody.
2. Relapse post-autologous transplant.
3. Relapse post-allogeneic transplant.

   d. Burkitt's Lymphoma

   i. Must have received Rituximab or another CD20 antibody in combination with anthracycline based chemotherapy regimen and have ONE of the following:

<!-- -->

1. Primary refractory lymphoma.
2. Relapse within 6 months.
3. For relapse >6 months, failure of two different chemotherapy regimens appropriate for their disease and be ineligible to receive autologous transplant.

   i. Relapse post-autologous transplant. ii. Relapse post-allogeneic transplant.
4. Able to provide written informed consent.
5. Negative urine or serum pregnancy test in females of childbearing potential at screening.
6. Willingness of women of reproductive potential and their partners to observe highly effective birth control methods for duration of treatment and for 1 month following the last dose if study treatment.
7. Karnofsky performance score ≥70.
8. Expected survival >12 weeks.
9. Patient has demonstrated compliance with prior therapies.
10. Able to take oral medications.
11. Adequate coagulation, defined as activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) and prothrombin (PT) or (international normalized ratio (INR) not greater than 1.5 x upper limit of normal (ULN).
12. Patients are required to have the following washout periods prior to planned Cycle 1 Day 1 (C1D1). In addition, prior treatment-related adverse events (AEs) must have recovered to Grade ≤ 1 with the exception of alopecia and Grade 2 peripheral neuropathy.

    1. Targeted agents, investigational agents, therapeutic monoclonal antibodies or cytotoxic chemotherapy: 5 half-lives or 2 weeks, whichever is shorter.
    2. immunoconjugated antibody treatment within 10 weeks prior to randomization.
    3. broad field radiation (≥ 30% of the bone marrow or whole brain radiotherapy) must be completed 14 days prior to study enrollment.
    4. palliative limited field radiation must be completed 7 days prior to study enrollment.

Inclusion Criteria to START Pirtobrutinib Bridging:

1. Absolute neutrophil count (ANC) ≥1000 with no G-CSF within 7 days or pegylated G-CSF within 14 days unless patient has biopsy proven bone marrow involvement.
2. Platelets≥50,000 with no transfusion within 7 days unless patient has biopsy proven bone marrow involvement.
3. Hemoglobin ≥8g/dL (≥80 g/L) [blood transfusions are allowable to reach this goal].
4. Adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine transaminase (ALT) <3 x upper limit of normal (ULN) or < 5 x ULN with documented liver involvement; serum bilirubin <1.5 x ULN or <3 x ULN with documented liver involvement , or considered not clinically significant as per the clinical PIs discretion (e.g. Gilbert's or indirect hyperbilirubinemia) or felt to be due to underlying disease.
5. Adequate renal function, defined as creatinine clearance≥50 ml/min.

   1. No IV hydration within 24 hours of eligibility.
   2. No dialysis dependent renal failure.

Inclusion criteria for Pirtobrutinib Maintenance (part B)

1. Recovery of neutrophils count after CAR T-cell infusion with ANC ≥1000/dL without G-CSF within the last 7 days.
2. Recovery of platelet count after CAR T-cell infusion with platelet count ≥50,000/dL.
3. Adequate hepatic function, defined as back to baseline or AST and ALT <3 x upper limit of normal (ULN); serum bilirubin and alkaline phosphatase <3 x ULN, or considered not clinically significant as per the clinical PI's discretion (e.g., Gilbert's or indirect hyperbilirubinemia) or felt to be due to underlying disease.
4. Adequate renal function, defined as creatinine clearance≥40 ml/min.
5. Evidence of response or stable disease (complete response/partial response/stable disease) at day 28 after CAR T-cell therapy.

Inclusion Criteria for Apheresis and LV20.19 CAR T-cells:

1. Active Measurable disease must be documented within 4 weeks of lymphodepletion start defined as nodal lesions greater than 15 mm in the long axis or extranodal lesions >10 mm in long and short axis OR bone marrow involvement that is biopsy proven for B-cell NHL.
2. Absolute cluster of differentiation (CD) 3 count≥50 mm^3.
3. MRI brain and Lumbar Puncture with cerebrospinal fluid (CSF) analysis by cytology and flow cytometry without evidence of central nervous system (CNS) involvement ONLY in patients with history of CNS involvement or clinical suspicion at the time of enrollment.
4. Adequate cardiac function as indicated by New York Heart Association (NYHA) classification I or II AND left ventricular ejection fraction of ≥45% (by echocardiogram (ECHO) or MUGA) and adequate pulmonary function as indicated by room air oxygen saturation of ≥92%.
5. No contraindication to central line access.
6. ANC≥1000 with no pegylated G-CSF within 14 days unless patient has biopsy proven bone marrow involvement.
7. Platelets≥50,000 with no transfusion within 72 hours unless patient has biopsy proven bone marrow involvement.
8. Adequate hepatic function, defined as AST and ALT <3 x upper limit of normal (ULN); serum bilirubin and alkaline phosphatase <3 x ULN, or considered not clinically significant as per the clinical PIs discretion (e.g. Gilbert's or indirect hyperbilirubinemia) or felt to be due to underlying disease.
9. Adequate renal function, defined as creatinine clearance≥50 ml/min. a. No IV hydration within 24 hours of eligibility. b. No dialysis dependent renal failure.

Exclusion Criteria:

A potential subject who meets any of the following exclusion criteria is ineligible to participate in the study.

1. Positive beta-human chorionic gonadotropin (HCG) in female of child-bearing potential or plan to become pregnant during the study or within 1 month of the last dose of study treatment and women who are current lactating or plan to breastfeed during the study or within 1 week of the last dose of study treatment.
2. Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection based on criteria below:

   1. HBV: Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation before randomization. Patients who are hepatitis B PCR positive will be excluded.
   2. Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before randomization. Patients who are hepatitis C RNA positive will be excluded.
3. Known active cytomegalovirus (CMV) infection (Unknown or negative status are eligible).
4. History of significant autoimmune disease OR active, uncontrolled autoimmune phenomenon requiring steroid therapy defined as >20 mg of prednisone or equivalent daily.
5. Presence of ≥ grade 3 non-hematologic toxicities as per CTCAE version 5.0 from any previous treatment unless it is felt to be due to underlying disease.
6. Concurrent use of investigational therapeutic agents or enrollment on another therapeutic clinical trial at any institution. Minimum of 14 days or 5 half-lives of the drug (whichever is shorter) washout prior to apheresis.
7. Refusal to participate in the long-term follow-up protocol.
8. Patients with active CNS involvement by malignancy on MRI or by lumbar puncture.

   1. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment and a remission documented within 8 weeks of planned CAR-T cell infusion by MRI brain and CSF analysis.
9. Previous recipients of allogeneic hematopoietic stem cell transplantation (AHCT) are excluded if they are <100 days post-transplant, have evidence of active graft-versus-host-disease (GVHD) of any grade, or are currently on immunosuppression.
10. Prior allogeneic CAR T-cell therapy <100 days from prior CAR T-cell treatment.
11. Previous recipients of autologous CAR-T cell therapy directed at either cluster of differentiation 19 (CD19) or CD20 are excluded if they are <100 days post prior CAR-T cell treatment (does not include re-enrollment) or have >5% residual circulating CAR-T as measured by flow cytometry using a CD19 CAR detection reagent (Miltenyi Biotec).

    a. Patients with prior CAR-T treatment against CD19 or CD20 must have repeat biopsy post-CAR-T cell therapy confirming a minimum of 5% CD19 or CD20 positivity by immunohistochemistry or flow cytometry.
12. Anti-CD20 antibody treatment within 4 weeks of cell infusion.
13. Anti-CD19 antibody treatment within 4 weeks of cell infusion.
14. Cytotoxic chemotherapy treatment within 14 days or steroid treatment (other than replacement dose steroids) within 7 days prior to apheresis collection for CAR-T cells.
15. No other oral chemotherapeutic agents or antibody directed treatment after starting pirtobrutinib other than steroids or radiation to a single site in a palliative fashion.
16. Patients post solid organ transplant who develop high grade lymphomas or leukemias.
17. Concurrent active malignancy other than basal or squamous cell carcinomas of the skin (underlying low-grade lymphoma chronic lymphocytic leukemia/Follicular lymphoma (FL) / Marginal zone lymphoma (MZL) is allowable in patients with transformed large cell lymphoma/Richter's.
18. Patients who experienced a major bleeding event or grade ≥ 3 arrhythmia on prior treatment with a BTK inhibitor.
19. History of stroke or intracranial hemorrhage within 6 months of randomization.
20. Significant cardiovascular disease defined as myocardial infarction within 6 months of randomization, congestive heart failure with ejection fraction <30%, active unstable angina, QT prolongation (QTcF)>470 msec on ECG.
21. Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of the study drug.
22. Patients requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist.
23. Patients who had surgery within 4 weeks prior to randomization.
24. Patients who have received vaccination with live vaccine within 28 days prior to randomization.
25. Patients with known hypersensitivity to any of the excipients of pirtobrutinib.

    Special Criteria Regarding Fertility and Contraception

    Female subjects of reproductive potential (women who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone a sterilization procedure [hysterectomy or bilateral oophorectomy]) must have a negative serum or urine pregnancy test performed at screening.

    Due to the high-risk level of this study, while enrolled, all subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). Additionally, if participating in sexual activity that could lead to pregnancy, the study subject must agree to use reliable and double barrier methods of contraception during the follow-up period of the protocol.

    Acceptable birth control includes a combination of two of the following methods:

    • Combined estrogen and progestin containing hormonal contraception associated with inhibition of ovulation given orally, intravaginally, or transdermally

    • Progestin-only hormonal contraception associated with inhibition of ovulation given orally, by injection, or by implant

    • Intrauterine device (IUD)

    • Intrauterine hormone-releasing system (IUS)

    • Vasectomized partner

    • Sexual abstinence: considered a highly effective method only if defined as refraining from heterosexual intercourse during an entire period of risk associated with the study treatment. The reliability of sexual abstinence will be evaluated in relation to the duration of the study and to the usual lifestyles of the patient.

    • Female sterilization

    • Fallopian tube implants (if confirmed by hysterosalpingogram) Oocyte donation is prohibited during the duration of participation on this protocol and for 1 month after the last dose of study drug.

    Subjects who are not of reproductive potential (women who are premenarche or have been post-menopausal for at least 24 consecutive months which is non-therapy induced or have undergone hysterectomy tubal ligation, salpingectomy, and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraception.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events After CAR 20/19-T Cell Infusion | Up until 28 days after infusion
  This measure is the number of adverse events with grade 3 to 5 severity per Common Terminology Criteria for Adverse Events (ver. 5) occurring during the first 28 days following infusion.
Number of Adverse Events After Pirtobrutinib Administration in Part A | 14 days prior to apheresis until the start of lymphodepletion
  Pirtobrutinib will be administered at 200 mg/day orally starting at least 14 days prior to apheresis as bridging until the start of lymphodepletion. This measure is the number of adverse events with grade 3 to 5 severity per Common Terminology Criteria for Adverse Events (ver. 5).
Number of Adverse Events After Pirtobrutinib Administration in Part B | Day 28 until up to one year
  Pirtobrutinib will be started again at 200 mg/day orally on day 28-120 for up to one year as maintenance post cell infusion. This measure is the number of adverse events with grade 3 to 5 severity per Common Terminology Criteria for Adverse Events (ver. 5).

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Shah, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No